CLINICAL TRIAL: NCT03992690
Title: Training With Brain-machine Interfaces, Visuo-tactile Feedback and Assisted Locomotion for Patients With Chronic Complete Paraplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: the Alberto Santos Dumont Association for Research Support (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XW-[2019]-023
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Chronic Paraplegia
MeSH Terms: interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WANR protocol (Experimental): Including training with Brain-machine interfaces, visuo-tactile feedback and assisted locomotion
  Interventions: Device: Brain-machine Interfaces, Visuo-tactile Feedback and Assisted Locomotion, or the WANR protocol
- Classical physiotherapy protocol (Active Comparator): Training with classical physiotherapy protocol
  Interventions: Device: Training with traditional physiotherapy protocol

INTERVENTIONS:
Device: Brain-machine Interfaces, Visuo-tactile Feedback and Assisted Locomotion, or the WANR protocol — Training integrating virtual-reality avatar driven by a brain-machine interface, with tactile feedback through patient's forearms, and assisted locomotion, for neurorehabilitation of SCI patients.
  Arms: WANR protocol
Device: Training with traditional physiotherapy protocol — Stretching
  Arms: Classical physiotherapy protocol

SUMMARY:
The purpose of this research is to compare the effectiveness of a training protocol integrating Brain-machine Interfaces, Visuo-tactile feedback and Assisted Locomotion (referred to as the Walk Again Neurorehabilitation protocol, or WANR), with classical physiotherapy training for patients with chronic complete paraplegia due to spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* 1. Discomplete spinal cord injury;
* 2. Traumatic etiology;
* 3. American Spinal Injury Association Impairment Scale(ASIA) A grade;
* 4. The level of SCI in T9-T12;
* 5. ≥12 months post injury;
* 6. Considered independents to perform daily life activities: feeding, dressing, capability with wheelchair;
* 7. Emotional stability;

Exclusion Criteria:

* 1. Absence of SCI, or presence of multi-segmental injury;
* 2. SCI non-traumatic etiology;
* 3. Age<18 years or Age>60 years;
* 4. Emotional instability;
* 5. Unavailable time to join the protocol activities;
* 6. Already enrolled in other research protocol;
* 7. Acute or chronic decompensated comorbidities (e.g. Hypertension, Diabetes, cardiomyopathy, chronic respiratory insufficiency, chronic renal insufficiency, hepatopathy, or any other neurological disorders besides the SCI);
* 8. Alcohol/drugs abuse and dependence;
* 9. Psychiatric disorders (exception: treated depression);
* 10.Cognitive deficit; visual deficit; auditory deficit;
* 11. Incapacitating pain;
* 12. Pregnancy;
* 13. Presence of limb amputations (exception: hand distal phalanges);
* 14. Peripheral neuropathy associated (e.g.: brachial plexus injury, carpal tunnel syndrome);
* 15. Muscle injury associated (e.g. myotendinous rupture, burning injury, muscle-compartment syndrome);
* 16. Neuromuscular disease associated (ex: myopathy) or lower limb fractures within the past six months;
* 17. Movement disorders(e.g. ataxia);
* 18. Use of medication that can negatively impact on neurological/motor recovery;
* 19. Presence of joint deformities, presence of fractures;
* 20. Lower limb spasticity MAS (Modified Ashworth Scale)>2;
* 21. Pressure ulcer: considering grade 3 or 4, injury size and body location;
* 22. Cephalic metallic /magnetic implants (exception: MRI compatible implants);
* 23. Presence of cardiac or neural pacemaker;
* 24. Use of devices/tubes: tracheostomy, gastrostomy, nasogastric, long-term bladder catheterization, cystostomy, colostomy, totally implanted catheter system, arteriovenous dialysis fistula;
* 25. Severe osteoporosis (Tscore>-4);
* 26. Syringomyelia;
* 27. Lokomat or ZeroG training within the prior 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of Lower limbs Motor function: ASIA motor score (LEMS) at the ending time point | After nine-months of training
  The LEMS evaluates motor function on a scale of 0 (no motor function) to 5 (full motor function) for 5 lower extremity muscle groups with a 50-point maximum (25 per side)

SECONDARY OUTCOMES:
The change of nociception improvement: ASIA pin-prick sensory score | After nine-months of training
  Testing of a key point in each of the 28 dermatomes (from C2 to S4-5) on the right and left sides of the body that can be readily located in relation to bony anatomical landmarks. At each of these key points, sensation of pin prick is examined:
  Appreciation of pin prick sensation at each of the key points is separately scored on a three-point scale, with comparison to the sensation on the patients' cheek as a normal frame of reference:
  0 = absent
  1= altered (impaired or partial appreciation, including hyperesthesia)
  2 = normal or intact (similar as on the cheek)
  NT = not testable
  The maximum scale is 112
Improvement of Walking index for SCI (WISCI) | After nine-months of training
  The subject is observed by the trained personnel and the WISCI level is recorded on the scale of 0 to 20 at baseline (Baseline WISCI). The subject is observed again at the defined interval (Interval WISCI). The change in score is calculated by subtracting the baseline WISCI from the Interval WISCI, which equals the change in WISCI (Changed WISCI).
Change of WHO-QoL bref | After nine-months of training
  The WHOQOL-BREF questionnaire contains two items from the Overall QOL and General Health and 24 items of satisfaction that divided into four domains. Raw domain scores for the WHOQOL were transformed to a 4-20 score according to guidelines
Change of post-void residual urine | After nine-months of training
  Usually, the value is less than 50 ml. A post-void residual urine greater than 50 ml is a significant amount of urine and increases the potential for recurring urinary tract infections. In adults older than 60 years, 50-100 ml of residual urine may remain after each voiding because of the decreased contractility of the detrusor muscle

CONTACTS AND LOCATIONS:
Overall Officials: Guo-Guang Zhao, M.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided